CLINICAL TRIAL: NCT00703560
Title: Molecular Basis of Interferon Response in HCV
Brief Title: Study of Hepatitis C Virus (HCV) Viral Kinetics in HIV/HCV and HCV Patients
Acronym: VK
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Mamta Jain, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: 102005-009; K23AI065630 (NIH)
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Hepatitis C
Keywords: HCV; Genotype 1; HIV co-infection; viral kinetics; HCV quasi-species; Hepatitis C genotype 1; HIV Infections
MeSH Terms: conditions — Hepatitis C; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: HIV and HCV genotype 1 coinfected (any race)
- 2: HCV genotype 1 (any race)

SUMMARY:
The purpose of this study is to evaluate what happens to hepatitis C virus in response to treatment with pegylated interferon and ribavirin in patients with HCV compared to those with HIV and HCV.

This research is being done to help us identify how the composition of HCV changes with interferon in different populations. We will examine how quickly HCV is cleared from your body and what factors may influence that clearance. This information may help us find better treatments for HCV.

DETAILED DESCRIPTION:
All patients who participate in this study will have frequent blood drawn in order to measure how quickly HCV virus declines. Pegylated interferon and ribavirin are not provided by the study, but will be obtained as part of standard of care treatment for hepatitis C. Participants must be willing to spend 48 hours in the hospital for frequent blood draws. They will be compensated for their time.

All patients must be HCV genotype 1. All patients must have a liver biopsy prior to enrollment into study. (This is not provided by the study).

HIV-infected patients must have a CD4 cell count>300. If HIV-infected and on antiretroviral therapy for HIV, they must be on a stable regimen for 12 weeks. The HIV regimen can not include didanosine (Videx).

ELIGIBILITY:
Inclusion Criteria:

1. HCV infection, as documented by the presence of circulating levels of HCV RNA by any RT-PCR or bDNA assay performed by a laboratory with a CLIA certification or its equivalent within 52 weeks prior to study entry.
2. HCV RNA >1000 IU/ml.
3. Documented genotype 1 performed by any CLIA certified lab.
4. Men and women age 18 to 65 years.
5. Ability and willingness of subject or legal guardian/representative to give written informed consent.
6. Female study volunteers of reproductive potential must be willing to use two methods of birth control in order to prevent pregnancy while on IFN/RBV.

For HIV infected patients:

1. HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
2. CD4+ cell count ³ 300 cells/mm3 within the prior 12 weeks at a CLIA certified lab or its equivalent.
3. Subject may be HAART naïve, but if on HAART should be on a stable regimen for 12 weeks The HAART regimen cannot include didanosine (Videx). Interaction with ribavirin and didanosine has led to fatal hyperlactatemia in a few patients.

Exclusion Criteria:

1. Unwilling to be admitted for 48 hours for serial blood draws for virology studies.
2. Hepatitis B surface antigen (HBsAg) positivity.
3. Prior IFN -based therapy.

Additional Exclusion for HIV-infected:

1. Current symptomatic HIV disease (i.e., AIDS-defining illnesses).
2. HAART regimen that contains Videx (Didanosine). Subject may previously have been on didanosine but if on a new HAART regimen should be on the regimen for 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCV genotype 1 with or without HIV-infection of any race.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2005-09; Primary Completion 2011-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Comparison of interferon effectiveness (as measured by epsilon) in HIV/HCV to HCV alone and African American to Caucasians. | 72 weeks

SECONDARY OUTCOMES:
SVR rate in HIV/HCV vs. HCV and African Americans vs. Caucasians | 72 weeks
Comparison of HCV quasi-species diversity | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mamta K. Jain, MD, MPH, Principal Investigator — University of Texas Southwestern Medical Center

REFERENCES:
- [Derived] Jain MK, Pasipanodya JG, Alder L, Lee WM, Gumbo T. Pegylated interferon fractal pharmacokinetics: individualized dosing for hepatitis C virus infection. Antimicrob Agents Chemother. 2013 Mar;57(3):1115-20. doi: 10.1128/AAC.02208-12. Epub 2012 Nov 26. PMID 23183434